CLINICAL TRIAL: NCT00005095
Title: Northwestern Ovarian Cancer Early Detection & Prevention Program: A Specimen and Data Study
Brief Title: Specimen and Data Study for Ovarian Cancer Early Detection and Prevention
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lee Shulman, Professor, Northwestern University
Other Study IDs: NU 99G8; P30CA060553 (NIH); NU-99G8 (Other: Northwestern University IRB); NCI-G00-1753 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2); Ovarian Cancer; Sarcoma; Uterine Leiomyomata; Vaginal Cancer; Vulvar Cancer
Keywords: ovarian epithelial cancer; hereditary breast/ovarian cancer (BRCA1, BRCA2); fallopian tube cancer; ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; endometrial cancer; uterine sarcoma; vaginal cancer; cervical cancer; vulvar cancer; uterine leiomyomata
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome; Ovarian Neoplasms; Sarcoma; Myofibroma; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial | interventions — CA-125 Antigen; Surveys and Questionnaires; Surgical Procedures, Operative; Buthionine Sulfoximine; Hysterectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subject's blood and other specimens are collected their follow-up clinic appointments, as needed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High Risk for Ovarian Cancer: Women who are at increased risk of ovarian cancer based on family or personal medical history who are participating in the Northwestern Ovarian Cancer Early Detection and Prevention Program clinic.
  Interventions: Other: Ca-125; Other: screening questionnaire administration; Procedure: Surgery
- Suspected or diagnosed gynecological condition: Women who are planning to undergo surgery for their gynecological condition
- Control Group: Healthy subjects with no history of cancer and at general risk.

INTERVENTIONS:
Other: Ca-125 — Subject's blood collected at their follow-up blood draw will be assessed for biomarkers that could lead to a panel for detecting early stage ovarian cancer.
  Groups: High Risk for Ovarian Cancer
Other: screening questionnaire administration — Questionnaires designed to assess quality of life for women at increased risk of ovarian cancer will be administered to the subjects. Clinical data will also be collected.
  Other Names: Questionnaire
  Groups: High Risk for Ovarian Cancer
Procedure: Surgery — Subjects will be assessed for high risk factors.
  Other Names: BSO, fallopian tubes, TAH, hysterectomy, bilateral salpingectomy, STIC
  Groups: High Risk for Ovarian Cancer

SUMMARY:
RATIONALE: To improve strategies for detection and prevention of early-stage disease.

PURPOSE: This research study is collecting specimens and data to develop better methods for early detection and prevention of ovarian cancer among the high risk population and those who have the disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify and develop highly sensitive and specific tumor markers for the detection and management of ovarian cancer and other gynecological malignancies.
* To identify new prevention approaches and therapies.
* To identify measures to improve the quality of life for women at increased risk for developing the disease and for women diagnosed with ovarian cancer.

OUTLINE: Subjects undergo periodic specimen and data collection for research studies, including molecular, biochemical, functional, and genetic marker studies. Participants may have samples of blood, tissue, or body fluids (such as ascites, pleural fluid or urine), or any combination of the aforementioned samples obtained to develop tumor markers to detect early stage or recurrent ovarian cancer.

The results from the biomarker research studies will not be reported to the patient or the physician. In the future, if any of the experimental tumor markers are found to be effective in detecting early stage ovarian cancer, and the patient's result is abnormal, the patient and physician will be notified.

Subjects may be asked to complete a combination of questionnaires designed to evaluate psychological functioning among women enrolled in a comprehensive ovarian cancer early detection program who are at increased risk for developing disease as compared to women currently diagnosed with ovarian cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Considered to be at increased risk for developing ovarian cancer, as defined by one of the following:

    * Has at least one first-degree relative (mother, sister, or daughter) with ovarian, primary peritoneal, or fallopian tube cancer
    * Has at least two first or second degree relatives diagnosed before age 50 with either ovarian, primary peritoneal, fallopian tube, and/or pancreatic cancer who have tested positive for hereditary cancer syndrome that includes an increased risk of gynecologic cancer (e.g., BRCA1/2 or Lynch Syndrome)or have increased risk as deemed by a certified genetic counselor
    * A personal or family history of a hereditary cancer syndrome that includes an increased risk of gynecologic cancer
    * Increased risk as deemed by a certified genetic counselor
  * Undergoing surgery for a gynecologic condition, including any of the following:

    * Diagnosis of a reproductive cancer
    * Benign gynecological condition (e.g., uterine leiomyomata, endometriosis, pelvic inflammatory disease, or follicular or corpus luteum ovarian cysts)
    * Highly suspicious adnexal mass
    * Risk-reducing prophylactic oophorectomy

PATIENT CHARACTERISTICS:

Age

* Between the ages of 18 and 80

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women at high risk of ovarian cancer due to family or personal medical history, or a gynecologic abnormality.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2000-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
The development of ultrasound and serum tumor markers for the detection and management of ovarian cancer and other | 1 year
  To identify markers to allow for presymptomatic testing for ovarian and other gynecological malignancies

SECONDARY OUTCOMES:
new prevention approaches and therapies for risk assessment | 1 year
  To identify new prevention approaches and therapies by researching and reviewing the risk of developing disease.
The develop of measures to improve the quality of life for women at increased risk for developing the disease and for women diagnosed with ovarian cancer | 1 year
  To identify the measurements to improve the quality of life for women at increased risk for developing the disease

CONTACTS AND LOCATIONS:
Overall Officials: Lee P. Shulman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- See also: Ovarian, Fallopian Tube, and Primary Peritoneal Cancer Research — https://www.cancer.gov/types/ovarian/research